CLINICAL TRIAL: NCT03379948
Title: Central and Peripheral Venous Catheters Associated Blood Stream Infection in the Critically Ill Patients in Assiut University Hospital
Brief Title: Central and Peripheral Venous Catheters Associated Blood Stream Infection in ICU in Assiut University
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Nassar Abd El Hameed Ali, principal investigator, Assiut University
Other Study IDs: CAPVCABSIITCIPIAUH
Record Dates: First submitted 2017-12-16; First posted 2017-12-20 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Blood Stream Infection
MeSH Terms: interventions — Blood Culture; Blood Cell Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 with central venous line: lab investigation Complete blood count blood culture
  Interventions: Diagnostic Test: blood culture
- Group 2 with only peripheral line: lab investigation Complete blood count blood culture
  Interventions: Diagnostic Test: blood culture

INTERVENTIONS:
Diagnostic Test: blood culture — blood culture to diagnose blood stream infection
  Other Names: complete blood count

SUMMARY:
Catheter related infections (CRIs) were found to be associated with several risk factors, including patient related risk factors such as age, gender, clinical status and catheter related risk factors such as the vascular access location, dwelling time, catheter type and number of lumens. In addition to the inserted solution type and the experience of the professional who performs the procedure ,These factors constitute important strategic points for actions to compare the infectious complications of peripheral versus central venous catheters in critically ill patients.

DETAILED DESCRIPTION:
Nosocomial (hospital-acquired) bloodstream infections (BSIs) are an important cause of morbidity and mortality, with an estimated 250,000 cases occurring each year in the United States.

BSIs may be either primary or secondary. Secondary infections are related to infections at other sites, such as the urinary tract, lung, postoperative wounds, and skin. Most nosocomial BSIs are primary, as illustrated by the United States Centers for Disease Control and Prevention's National Nosocomial Infection Surveillance system, in which 64 percent of the nosocomial BSIs reported were primary BSIs. While some primary BSIs have no identifiable source, most are associated with intravascular catheters, and central venous catheters (CVCs) in particular.

Critically ill patients require intravenous administration of fluids and drugs.This can be achieved via peripheral or central catheters. Each device is associated with both mechanical and infectious complications. Complications associated with central lines are judged to be more severe. Some patients actually require the insertion of a central line due to the venous toxicity of the drugs or to the necessity of making sure that the infusion is regularly administered (example: high dose catecholamine infusion). Some physicians believe that most Intensive Care Unit (ICU) patients should have a central venous line inserted, whereas others feel that some patients may receive active drugs via a peripheral line in selected instances.

Endpoints are the rate of mechanical complications (difficulty in inserting the line, need for repeat insertion attempts, occurrence of arterial puncture, occurrence of pneumothorax) and of infectious complications (local catheter infection or catheter-related bloodstream infection).

ELIGIBILITY:
Inclusion Criteria:

* All patient at ICU Diagnosed nosocomial infection

Exclusion Criteria:

* Patients exist already infected before admission at hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presented to assiut university hospital admitted at intensive care unit
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
compare the infectious complications of peripheral versus central venous catheters in critically ill patients | 7 days
  by blood sample

CONTACTS AND LOCATIONS:
Overall Officials: mohamed maghraby, MD, Study Chair — ASSIUT UNIVERSTAY
Locations (1):
- Assiut Universtay Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
i wiil share it

REFERENCES:
- [Background] Chen HS, Wang FD, Lin M, Lin YC, Huang LJ, Liu CY. Risk factors for central venous catheter-related infections in general surgery. J Microbiol Immunol Infect. 2006 Jun;39(3):231-6. PMID 16783454
- [Background] Timsit JF. [Updating of the 12th consensus conference of the Societe de Reanimation de langue francaise (SRLF): catheter related infections in the intensive care unit]. Ann Fr Anesth Reanim. 2005 Mar;24(3):315-22. doi: 10.1016/j.annfar.2004.12.022. French. PMID 15792575
- [Background] Holton D, Paton S, Conly J, Embree J, Taylor G, Thompson W. Central venous catheter-associated bloodstream infections occurring in Canadian intensive care units: A six-month cohort study. Can J Infect Dis Med Microbiol. 2006 May;17(3):169-76. doi: 10.1155/2006/781735. PMID 18418495
- [Background] Lorente L, Henry C, Martin MM, Jimenez A, Mora ML. Central venous catheter-related infection in a prospective and observational study of 2,595 catheters. Crit Care. 2005;9(6):R631-5. doi: 10.1186/cc3824. Epub 2005 Sep 28. PMID 16280064